CLINICAL TRIAL: NCT02142387
Title: Clinical Effects of a New Dispatcher-Assisted Basic Life Support Training Program in a Metropolitan City: A Before-and-After Intervention Study
Brief Title: Effects of a New Dispatcher-Assisted Basic Life Support Training Program
Acronym: HEROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Do Shin, professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-heros-01
Record Dates: First submitted 2014-05-13; First posted 2014-05-20 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Out of Hospital Cardiac Arrest
Keywords: cardiac arrest; dispatcher-assisted bystander cardiopulmonary resuscitation; survival
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New DA-BLS training program (Active Comparator): A one-hour training course that includes a 30-minute video-based self-instruction (VSI) training session, a short role-play, and a debriefing. The video consists of a bystander CPR simulation with dispatcher instructions using the trainee's own phone and practice session following demonstration by a simulated layperson. After watching the video clip, all trainees are divided into two groups and conduct a role-play as dispatchers and laypersons for 15 minutes. Finally, there is a 15-minute debriefing session with several assignments. The HEROS program focuses on cooperation with a dispatcher, from recognition of cardiac arrest to performing DA-CPR, with hands-on practice so that laypersons can provide bystander CPR immediately in a real situation. Moreover, the HEROS program emphasizes practice for providing the correct address of the scene and switching to speakerphone mode, especially for the elderly.
  Interventions: Other: BLS CPR program with dispatcher assisted CPR simulation
- Current Basic Life Support (BLS) training program (No Intervention): A one-hour training program that was developed by the Korea Center for Disease Control and Prevention (CDC) and it was based on the American Heart Association (AHA) guideline (http://www.cdc.go.kr/board.es?mid=a20503050000&bid=0021&tag=&act=view&list_no=127655). The program consists of a 30-minute VSI, and a 30-minute practice debriefing session. It focuses on detailed techniques for performing high-quality chest compressions including the correct hands and body position of the bystanders.

INTERVENTIONS:
Other: BLS CPR program with dispatcher assisted CPR simulation — the training program more focuses on cooperation with a dispatcher, from recognition to perform DA-CPR and hands-on practice.
  Arms: New DA-BLS training program

SUMMARY:
Despite aggressive cardiopulmonary resuscitation (CPR) training, the outcome of cardiac arrest is not good. The problem is method of education. So, the investigators want to add the dispatcher-assisted CPR simulation into conventional CPR training. In this study, the study is aimed to investigate the effect of newer CPR training program.

DETAILED DESCRIPTION:
The training program focuses on working in team with dispatcher, performing all steps from recognizing cardiac arrest to performing CPR, together with the dispatcher. The one hours training session is split into four parts:

1. Video self-instruction manikin practice (30 min), including a brief introduction to automated external defibrillator (AED).
2. Practice in pairs (15 min). Practicing the dispatcher and rescuer role in a simulation to enhance learning.
3. Debriefing. Questions, answers and reflection (15 min).
4. Homework. Leaflet with tasks like learn how to activate the speaker function on your own phone.

The main difference between dispatcher-assisted basic life support (DA-BLS) and traditional BLS training is that DA-BLS provides the scenes and interactive experiences on calling emergency medical service (EMS) and receiving CPR instruction via telephone speaker function, following up the skill training by scenario simulation training.

ELIGIBILITY:
Inclusion Criteria:

* All out-of-hospital cardiac arrest (OHCA) patients with presumed cardiac etiology who are 19 years of age or older and assessed and treated by EMS providers after dispatched by the EMS dispatch center will be included.

Exclusion Criteria:

* We will exclude patients with non-cardiac etiology, prolonged cardiac arrest with a suspected duration more than 30 minutes, cases such as livor mortis or rigor mortis, and decapitated or decomposed body, and patients who have "Do-Not-Resuscitate" card documented by doctor.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18822 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Do Shin, MD, MPH, PHD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park GJ, Song KJ, Shin SD, Hong KJ, Kim TH, Park YM, Kong J. Clinical effects of a new dispatcher-assisted basic life support training program in a metropolitan city. Medicine (Baltimore). 2022 Jul 15;101(28):e29298. doi: 10.1097/MD.0000000000029298. PMID 35839001

RESULTS

PARTICIPANT FLOW:
Groups:
- New DA-BLS Training Program: A one-hour training course that includes a 30-minute video-based self-instruction (VSI) training session, a short role-play, and a debriefing. The video consists of a bystander CPR simulation with dispatcher instructions using the trainee's own phone and practice session following demonstration by a simulated layperson. After watching the video clip, all trainees are divided into two groups and conduct a role-play as dispatchers and laypersons for 15 minutes. Finally, there is a 15-minute debriefing session with several assignments. The program focuses on cooperation with a dispatcher, from recognition of cardiac arrest to performing DA-CPR, with hands-on practice so that laypersons can provide bystander CPR immediately in a real situation.
- Current Basic Life Support (BLS) Training Program: A one-hour training program that was developed by the Korea Center for Disease and Prevention (CDC) and it was based on the American Heart Association (AHA) guideline (http://www.cdc.go.kr/board.es?mid=a20503050000&bid=0021&tag=&act=view&list_no=127655). The program consists of a 30-minute VSI, and a 30-minute practice debriefing session. It focuses on detailed techniques for performing high-quality chest compressions including the correct hands and body position of the bystanders.
Period: Overall Study
Arm/Group | New DA-BLS Training Program | Current Basic Life Support (BLS) Training Program
Started | 2551 (Out-of-hospital cardiac arrest (OHCA) patients with presumed cardiac etiology.) | 16271
Completed | 1486 (Limited to the case where OHCA occurred in the private place.) | 8641
Not Completed | 1065 | 7630
Not completed — <19 years old | 49 | 326
Not completed — non-cardiac etiology | 504 | 3431
Not completed — CPR not performed | 74 | 473
Not completed — witnessed by paramedic | 139 | 917
Not completed — incomplete data | 1 | 9
Not completed — occurred not at home | 298 | 2474

BASELINE CHARACTERISTICS:
Groups:
- Districts Which Implement New DA-BLS Training Program: A one-hour training course that includes a 30-minute video-based self-instruction (VSI) training session, a short role-play, and a debriefing. The video consists of a bystander CPR simulation with dispatcher instructions using the trainee's own phone and practice session following demonstration by a simulated layperson. After watching the video clip, all trainees are divided into two groups and conduct a role-play as dispatchers and laypersons for 15 minutes. Finally, there is a 15-minute debriefing session with several assignments. The HEROS program focuses on cooperation with a dispatcher, from recognition of cardiac arrest to performing DA-CPR, with hands-on practice so that laypersons can provide bystander CPR immediately in a real situation. Moreover, the HEROS program emphasizes practice for providing the correct address of the scene and switching to speakerphone mode, especially for the elderly.
- Districts Which Keep Current BLS Training Program: A one-hour training program that was developed by the Korea CDC and it was based on the AHA guideline (http://www.cdc.go.kr/board.es?mid=a20503050000&bid=0021&tag=&act=view&list_no=127655). The program consists of a 30-minute VSI, and a 30-minute practice debriefing session. It focuses on detailed techniques for performing high-quality chest compressions including the correct hands and body position of the bystanders.
- Total: Total of all reporting groups
Arm/Group | Districts Which Implement New DA-BLS Training Program | Districts Which Keep Current BLS Training Program | Total
Number analyzed (Participants) | 1486 | 8641 | 10127
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74 [62 to 82] | 74 [62 to 82] | 74 [62 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 623 | 3487 | 4110
  Male | 863 | 5154 | 6017
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1486 | 8641 | 10127
witnessed by laypersons [Count of Participants; unit: Participants] — Witnessed by layperson means that someone (not paramedic) found cardiac arrest patients on the scene.
  Participants | 681 | 3993 | 4674
DA-CPR [Count of Participants; unit: Participants] — Dispatcher-assisted CPR (DA-CPR), identifying cardiac arrest through key questions, and helping laypersons provide appropriate chest compression when laypersons call 119 when the patient collapsed on the scene.
  Participants | 1139 | 6717 | 7856
bystander CPR [Count of Participants; unit: Participants] — bystander CPR means that laypersons provide chest compression to the cardiac arrest patient until the paramedics arrive on the scene.
  Participants | 859 | 5281 | 6140
shockable rhythm [Count of Participants; unit: Participants] — Shockable rhythm means that cardiac rhythm which can be shocked using automated external defibrillator including ventricular fibrillation and pulseless ventricular tachycardia.
  Participants | 187 | 1080 | 1267
level of ED [Count of Participants; unit: Participants] — An emergency department (ED) is formally categorized into level I, level II, III, or above level by law. The level of an ED is based on its resources, and level I and II EDs should be staffed by emergency physicians.
  Participants
    Level 1 | 12 | 1086 | 1098
    Level 2 | 1276 | 6533 | 7809
    Level 3 | 198 | 1022 | 1220

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Surviving to Hospital Discharge
Description: The study end points are survival to hospital discharge. Survival to discharge will be measured as proportions of patients who were discharged from a hospital with their spontaneous circulation recovered. This information will be collected from medical record review.
Time Frame: from date of discharge, assessed up to 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Districts Which Implement Newer DA-BLS Training Program: the out of hospital cardiac arrest victims who were given bystander CPR by whom trained as newer dispatcher-assisted BLS training program, which more focuses on cooperation with a dispatcher, from recognition to perform DA-CPR and hands-on practice.
  BLS CPR program with dispatcher assisted CPR simulation: the training program more focuses on cooperation with a dispatcher, from recognition to perform DA-CPR and hands-on practice.
- Districts Which Keep Traditional BLS Training Program: Control group commonly uses a one-hour training program which was developed by the Korea CDC. It focuses on detailed techniques of performing high-quality chest compressions.
Arm/Group | Districts Which Implement Newer DA-BLS Training Program | Districts Which Keep Traditional BLS Training Program
Number analyzed (Participants) | 1486 | 8641
Participants | 85 | 551
Statistical Analysis 1: Comparison: Districts Which Implement Newer DA-BLS Training Program vs Districts Which Keep Traditional BLS Training Program; Test type: Other; p = 0.34, Chi-squared

2. Secondary Outcome: Number of Participants With Return of Spontaneous Circulation (ROSC)
Description: The return of spontaneous circulation will be measured as proportion of the patients who were recovered their circulation at emergency department. This information will be collected from the medical review.
Time Frame: from date of cardiac arrest occurred, assessed up to 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Districts Which Implement Newer DA-BLS Training Program | Districts Which Keep Traditional BLS Training Program
Number analyzed (Participants) | 1486 | 8641
Participants | 544 | 3118
Statistical Analysis 1: Comparison: Districts Which Implement Newer DA-BLS Training Program vs Districts Which Keep Traditional BLS Training Program; Test type: Other; p = 0.7, Chi-squared

3. Secondary Outcome: Number of Participants With Good Neurological Recovery
Description: The Cerebral Performance Categories (CPC) score will be used to measure neurological recovery status: CPC 1 (good cerebral performance), CPC 2 (moderate cerebral disability), CPC 3 (severe cerebral disability), CPC 4 (coma or vegetative state), CPC 5 (brain death).
  We defined the good neurological recovery as CPC 1 or CPC 2. This information will be collected from medical record review.
Time Frame: from date of discharge, assessed up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Districts Which Implement Newer DA-BLS Training Program | Districts Which Keep Traditional BLS Training Program
Number analyzed (Participants) | 1486 | 8641
Participants | 42 | 316
Statistical Analysis 1: Comparison: Districts Which Implement Newer DA-BLS Training Program vs Districts Which Keep Traditional BLS Training Program; Test type: Other; p = 0.11, Chi-squared

ADVERSE EVENTS:
Time Frame: from date of discharge, assessed up to 3 months
Description: 1,401 cardiac arrest patients are died in the districts which implement new DA-BLS Training program.
  8,090 cardiac arrest patients are died in the districts which keep current BLS Training program.
Groups:
- Newer DA-BLS Training Program: A 30-minute video-based self-instruction (VSI) training session, a short role-play, and a debriefing. The video consists of a bystander CPR simulation with dispatcher instructions using the trainee's own phone and practice session following demonstration by a simulated layperson. After watching the video clip, all trainees are divided into two groups and conduct a role-play as dispatchers and laypersons for 15 minutes. Finally, there is a 15-minute debriefing session with several assignments. The HEROS program focuses on cooperation with a dispatcher, from recognition of cardiac arrest to performing DA-CPR, with hands-on practice so that laypersons can provide bystander CPR immediately in a real situation. Moreover, the HEROS program emphasizes practice for providing the correct address of the scene and switching to speakerphone mode, especially for the elderly.
- Current BLS Training Program: A one-hour training program that was developed by the Korea CDC and it was based on the AHA BLS provider course (http://www.cdc.go.kr/board.es?mid=a20503050000&bid=0021&tag=&act=view&list_no=127655). The program consists of a 30-minute VSI, and a 30-minute practice debriefing session. It focuses on detailed techniques for performing high-quality chest compressions including the correct hands and body position of the bystanders.
Arm/Group | Newer DA-BLS Training Program | Current BLS Training Program
All-Cause Mortality (participants affected / at risk) | 1401/1486 | 8090/8641
Serious Adverse Events (participants affected / at risk) | 1401/1486 | 8090/8641
Other Adverse Events (participants affected / at risk) | 0/1486 | 0/8641
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Newer DA-BLS Training Program (N=1486) | Current BLS Training Program (N=8641)
death (Cardiac disorders) | 1401 | 8090

LIMITATIONS AND CAVEATS:
This new DA-BLS training program was only used in the community health center. And it was difficult to identify whether laypersons who had performed bystander CPR actually received this new program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT02142387/Prot_SAP_000.pdf